CLINICAL TRIAL: NCT01613729
Title: An Open-label, Randomized, Multi-centre, Phase IVb, Parallel Study Group to Compare the Efficacy and Safety of 5 mg and 10 mg Rosuvastatin
Brief Title: Efficacy and Safety Study of 5 mg and 10 mg Rosuvastatin
Acronym: Cor16
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: D16 Pharma & Biotec Ltd. (Industry)
Collaborators: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other); Dhaka Medical College (Other); National Institute of Cardiovascular Diseases (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: corestin/bd/2012-16
Record Dates: First submitted 2012-06-04; First posted 2012-06-07 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Dyslipidemia
Keywords: Dyslipidemia; Rosuvastatin; Efficacy; Safety
MeSH Terms: conditions — Dyslipidemias | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosuvastation 5 Initiator Arm (Active Comparator): These patients will start the study with Rosuvastatin 5 mg and then after 12 weks they will be switched to Rosuvastatin 10 mg.
  Interventions: Drug: Rosuvastatin 5 mg
- Rosuvastatin 10 initiator arm (Active Comparator): These patients will continue with Rosuvastatin 10 mg and after 12 weeks they will be switched to Rosuvastatin 5 mg
  Interventions: Drug: Rosuvastatin 10 mg

INTERVENTIONS:
Drug: Rosuvastatin 5 mg — Rosuvastatin 5 mg
  Arms: Rosuvastation 5 Initiator Arm
Drug: Rosuvastatin 10 mg
  Arms: Rosuvastatin 10 initiator arm

SUMMARY:
The primary objective of the study is to compare the efficacy of Rosuvastatin 5 mg once daily with Rosuvastatin 10 mg once daily by assessment of the number of patients with hypercholesterolemia reaching the LDL-C target goal of <100 mg/dL after 12 weeks of therapy.

DETAILED DESCRIPTION:
This study will observe the followings:

1. To compare the effect of 5 mg/10 mg Rosuvastatin by assessment of the number of patients reaching LDL-C target goal after 24 weeks of therapy.
2. To compare the effect of 12 weeks therapy with 5 mg/10 mg Rosuvastatin on change in LDL-C (compare change from baseline).
3. To investigate the effect of 12 weeks therapy with 10 mg Rosuvastatin on change in LDL-C (compare values week 0 vs. week 12).
4. To investigate the safety of Rosuvastatin in regards to liver enzyme change, kidney function and muscle toxicity.
5. To compare the effect of 12 weeks therapy with 5 mg/10 mg Rosuvastatin on change in TC, HDL-C, TG, LDL-C density and HbA1c (compare change from baseline).
6. To investigate the effect of 12 weeks therapy with 10 mg Rosuvastatin on change in TC, HDL-C, TG, LDL-C density and HbA1c (compare values week 0 vs. week 12).
7. To investigate the effect of 12 weeks therapy on change in microalbuminuria in each treatment group (compare change from baseline).
8. To investigate the effect of 12 weeks therapy on change in BMI (compare change from baseline).

   The effects of the dose increase and the dose decrease from weeks 12 to 24 will be evaluated as follows:
9. To investigate the change in LDL-C by increasing the dose from 5 mg to 10 mg (compare values week 12 vs. 24).
10. To investigate the change in LDL-C by decreasing the dose from 10 mg to 5 mg (compare values week 12 vs. 24).
11. To investigate the change in TC, HDL-C, TG, LDL-C density and HbA1c by increasing the dose from 5 mg to 10 mg (compare values week 12 vs. 24).
12. To investigate the change in TC, HDL-C, TG, LDL-C density and HbA1c by decreasing the dose from 10 mg to 5 mg (compare values week 12 vs. 24).

ELIGIBILITY:
Inclusion Criteria:

* Age 45 - 75 years
* LDL - C between 130 mg/dL and 250 mg/dL
* TG < 400 mg/dL
* HbA1c < 7%
* Written informed consent to participate in the trial

Exclusion Criteria:

* Known hypersensitivity or history of SAE with another HMG-CoA reductase inhibitor, in particular any history of myopathy
* Active liver disease/severe hepatic impairment
* Treatment with cyclosporin or any disallowed drug
* Patients with unstable angina pectoris

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Rosuvastatin 5 mg once daily with Rosuvastatin 10 mg once daily by assessment of the number of patients with hypercholesterolemia reaching the LDL-C target goal of <100 mg/dL after 12 weeks of therapy. | 24 weeks

SECONDARY OUTCOMES:
To compare the safety | 24 weeks
  To investigate the effect of 12 weeks therapy on change in microalbuminuria in each treatment group (compare change from baseline).
  To investigate the effect of 12 weeks therapy on change in BMI (compare change from baseline).
  The effects of the dose increase and the dose decrease from weeks 12 to 24 will be evaluated
  to investigate the safety of Rosuvastatin in regards to Liver enzyme change, kidney function and muscle toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Nazrul Islam, FCPS, Principal Investigator — Professor of Cardiology; Pinaki Bhattacharya, MBBS, Study Director — D16 Pharma & Biotec
Locations (1):
- BSMMU, Dhaka, Dhaka Division, Bangladesh